CLINICAL TRIAL: NCT01314807
Title: Systemic Consequences and Comorbidities in Mild/Moderate COPD, Time for Action!
Brief Title: Systemic Consequences and Comorbidities in Mild/Moderate Chronic Obstructive Pulmonary Disease (COPD), Time for Action!
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Thierry Troosters, Prof. Dr., KU Leuven
Other Study IDs: The Rainbow study
Record Dates: First submitted 2011-03-09; First posted 2011-03-15 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood, cholesterol, LDL, HDL, creatinine, fibrinogen, glucose, insuline, NTproBNP, CRP, Hba1C
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- patients with COPD: patients who were defined as COPD, based on post-bronchodilator spirometry (GOLD criteria). Patients will have at least 10 pack years
- smoking controls: patients with at least 10 pack years who have no COPD (based on post-bronchodilator spirometry)
- non-smoking controls: patients with < 1 pack year who have no COPD (based on post-bronchodilator spirometry)

SUMMARY:
The aim of this prospective case-control study is to investigate the prevalence, severity and incidence of systemic consequences in newly detected patients with mild and moderate Chronic obstructive pulmonary disease (COPD). Special attention will be paid to skeletal muscle dysfunction and physical inactivity as these factors are, together with smoking, potentially modifiable.

DETAILED DESCRIPTION:
Three groups will be included in this study:

* Patients with COPD (cases)
* Patients with smoking history but no COPD (smoking controls)
* Patients with no smoking history and no COPD (non-smoking controls)

An extensive test battery will be performed at baseline and after 3 years:

Clinical assessment (height, weight and blood pressure)*

Complete pulmonary function ((post-bronchodilator)spirometry + diffusion)*

Sputum Induction

Fasting venous blood sample (fasting glucose, cholesterol, triglycerides, inflammatory markers, creatinine, NT pro BNP, hemoglobin, testosterone, vitamin D)

Vascular screening (arterial stiffness - arterial stenosis - CIMT)

Muscle force (peripheral + respiratory)*

Functional exercise capacity (6 MWT)**

Maximal exercise capacity (incremental cycle test)**

Dexa scan (osteoporosis - body composition)

Spiral CT scan of the chest

RX thorax - RX lumbar

Questionnaires (MRC, CCQ, SF-36, EQ5D, HADS, Exacerbation, CATZ)**

Physical activity monitoring (sensewear armband)*

* test will be repeated every 6 months

** test will be repeated every year

!!!! Remark (26/9/2013) Based on the last data analyses, in contrast to our expectations, we concluded that the two groups with a smoking history, with or without COPD change in a similar way over time. The length of the study will therefore be prolonged with 3 more years (6 years in total).

After 3 years the patients with a smoking history will be evaluated yearly, unless they were hospitalized for >5 days. In that case we will sooner contact these patients in order to pick up comorbidities in these patients.!!!

ELIGIBILITY:
Inclusion Criteria:

* age 40-80 years old

cases: spirometry (post-bronchodilator) based diagnosis of COPD (GOLD criteria) + smoking history of at least 10 pack-years and active smoking behavior till at least 10 years from the moment of enrollment.

smoking controls: no COPD (spirometry based) + smoking history of at least 10 pack-years and active smoking behavior till at least 10 years from the moment of enrollment.

non-smoking controls: no COPD (spirometry based) + < 1 pack year

Exclusion Criteria:

* Respiratory disorder other than COPD
* α1-antitrypsin deficiency
* Known history of significant inflammatory disease other than COPD
* COPD exacerbation within 4 weeks prior to study
* Lung surgery
* Recent diagnosis of cancer
* Therapy with oral corticosteroids in the last 6 weeks
* Significant cardiovascular comorbidity
* Significant orthopedic/musculoskeletal problems

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population-based sample from the general population: random selected patients from the environment of Leuven (Nelson Study), and co-workers from the University Hospital of Leuven
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-06; Primary Completion 2014-06 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of risk factors to develop comorbidities (vascular dysfunction, osteoporosis, muscle wasting and metabolic syndrome) | baseline
  Common risk factors: smoking, COPD, physical inactivity (steps (per day)and moderate intense PA (min/day) and systemic inflammation (CRP, fibrinogen, IL-6, IL-8, TNF-alpha). Specific risk factors: vascular (atherosclerosis (mean IMT carotid arteries), arterial stenosis (ankle brachial index) and arterial stiffness (brachial ankle pulse wave velocity)), bone (osteopenia: T-score < -1 at lumbar spine/femoral neck/total femur), muscle (fat free mass index < 15/16(female/male) and respiratory/peripheral muscle weakness; < 80%predicted), metabolic (syndrome): definition by AHA
Incidence and worsening of risk factors to develop comorbidities (vascular dysfunction, osteoporosis, muscle wasting and metabolic syndrome) | 3 years
  Common risk factors: smoking, COPD, physical inactivity (steps (per day)and moderate intense PA (min/day) and systemic inflammation (CRP, fibrinogen, IL-6, IL-8, TNF-alpha). Specific risk factors: vascular (atherosclerosis (mean IMT carotid arteries), arterial stenosis (ankle brachial index) and arterial stiffness (brachial ankle pulse wave velocity)), bone (osteopenia: T-score < -1 at lumbar spine/femoral neck/total femur), muscle (fat free mass index < 15/16 (female/male) and respiratory/peripheral muscle weakness; < 80%predicted), metabolic (syndrome): definition by AHA

CONTACTS AND LOCATIONS:
Overall Officials: Wim Janssens, Prof, Principal Investigator — KU Leuven; Thierry Troosters, Prof, Principal Investigator — KU Leuven
Locations (1):
- University Hospital Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Rodrigues FM, Demeyer H, Loeckx M, Hornikx M, Van Remoortel H, Janssens W, Troosters T. Health status deterioration in subjects with mild to moderate airflow obstruction, a six years observational study. Respir Res. 2019 May 18;20(1):93. doi: 10.1186/s12931-019-1061-7. PMID 31103027
- [Derived] Van Remoortel H, Hornikx M, Langer D, Burtin C, Everaerts S, Verhamme P, Boonen S, Gosselink R, Decramer M, Troosters T, Janssens W. Risk factors and comorbidities in the preclinical stages of chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2014 Jan 1;189(1):30-8. doi: 10.1164/rccm.201307-1240OC. PMID 24219412